CLINICAL TRIAL: NCT01272908
Title: Rituximab Phase IIIb Open-label, Multi-centre Assessment of Safety and Effectiveness in Patients With RA Following an Inadequate Response to One Prior Anti-TNF Inhibitor (RESET)
Brief Title: A Study of MabThera (Rituximab) in Patients With Rheumatoid Arthritis Who Have Failed on One Prior Anti-TNF Therapy (RESET)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20381
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — 1000 mg intravenously on Days 1 and 15

SUMMARY:
This study will evaluate the safety and effectiveness of MabThera (rituximab) in patients with active rheumatoid arthritis who are receiving methotrexate, and who have a previous or current inadequate response to one prior anti-TNF therapy. All patients will receive MabThera 1000 mg as an intravenous infusion on days 1 and 15. After the initial study phase of 24 weeks, eligible patients may receive one re-treatment with MabThera. The anticipated time on study treatment is 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18-80 years of age
* Moderate to severe active rheumatoid arthritis
* Inadequate response to a single previous or current treatment with an anti-TNF agent
* Methotrexate for at least 12 weeks, at a stable dose over the past 4 weeks

Exclusion Criteria:

* Previous treatment with MabThera
* Use of an anti-TNF agent within past 8 weeks (4 in the case of etanercept)
* Concurrent treatment with any Disease Modifying Anti-Rheumatic Drug (DMARD) other than methotrexate
* Active infection, or history of serious or chronic infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-07-18 (Actual); Primary Completion 2009-03-12 (Actual); Study Completion 2009-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (32):
- Canada (20):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Hamilton, Ontario
  - Mississauga, Ontario
  - Nepean, Ontario
  - Ottawa, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Laval, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Saint-Eustache, Quebec
  - Sainte-Foy, Quebec
  - Sherbrooke, Quebec
  - Trois-Rivières, Quebec
- Sweden (12):
  - Borås
  - Falun
  - Gothenburg
  - Jönköping
  - Kalmar
  - Karlskrona
  - Luleå
  - Malmo
  - Oskarström
  - Skövde
  - Stockholm
  - Sundsvall

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab + Methotrexate (MTX): Participants received rituximab 1000 milligrams (mg) intravenously (IV) and methylprednisolone 100 mg IV on Days 1 and 15. Participants should have been receiving a stable dose (for at least 12 weeks prior to Screening) of MTX 10-25 mg per week (mg/week) and a stable dose of folate (greater than or equal to [≥]5 mg/week) given as either a single weekly dose or as divided daily doses (per investigator discretion). Participants who, in the opinion of the investigator, achieved a clinically relevant response (Disease Activity Score based on 28-Joint Count [DAS28] score of greater than or equal to [≥]2.6) to the first course of treatment received one additional course of re-treatment with rituximab (2 IV infusions of rituximab 1000 mg [and methylprednisolone 100 mg], given 14 days apart), at any time between Week 24 and 48.
Period: Initial Treatment Period
Arm/Group | Rituximab + Methotrexate (MTX)
Started | 120
Completed | 112
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 5
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Period: Re-Treatment Period
Arm/Group | Rituximab + Methotrexate (MTX)
Started | 77 (Only participants with active disease as characterized by DAS-28 score ≥2.6 were included.)
Completed | 71
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: all participants who recieved any amount of infused medication whether or not they completed any further assessment.
Groups:
- Rituximab + MTX: Participants received rituximab 1000 mg IV and methylprednisolone 100 mg IV on Days 1 and 15. Participants should have been receiving a stable dose (for at least 12 weeks prior to Screening) of MTX 10-25 mg/week and a stable dose of folate (≥5 mg/week) given as either a single weekly dose or as divided daily doses (per investigator discretion). Participants who, in the opinion of the investigator, achieved a clinically relevant response (DAS28 score of ≥2.6) to the first course of treatment received one additional course of re-treatment with rituximab (2 IV infusions of rituximab 1000 mg [and methylprednisolone 100 mg] given 14 days apart), at any time between Week 24 and 48.
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events During the Initial Treatment Period - Overall Summary
Description: Percentage of participants who reported an AE or serious AE (SAE), a drug-related AE, who had an acute infusion reaction, an AE leading to study drug discontinuation, with an infection or serious infection, or who died.
Time Frame: Days 1, 2, 15, and 16 and Week 48 of Initial treatment period
Population: ITT Population
Measure: Number; unit: percentage of participants
Groups:
- Initial Treatment Period: Rituximab + MTX: Participants received rituximab 1000 mg IV and methylprednisolone 100 mg IV on Days 1 and 15. Participants should have been receiving a stable dose (for at least 12 weeks prior to Screening) of MTX 10-25 mg/week and a stable dose of folate (≥5 mg/week) given as either a single weekly dose or as divided daily doses (per investigator discretion).
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
percentage of participants
  With an AE | 85.0
  With a drug-related AE | 41.7
  With an acute infusion reaction | 20.8
  With AE leading to study drug discontinuation | 4.2
  With an SAE | 10.0
  With infections | 47.5
  With a serious infections | 2.5
  Who died | 0

2. Secondary Outcome: Percentage of Participants With Adverse Events During the Re-Treatment Period - Overall Summary
Description: Percentage of participants who reported an AE or SAE, a drug-related AE, who had an acute infusion reaction, an AE leading to study drug discontinuation, with an infection or serious infection, or who died.
Time Frame: Days 1, 2, 15, and 16 and Week 48 of Re-treatment period
Population: ITT Population
Measure: Number; unit: percentage of participants
Groups:
- Re-Treatment Period: Rituximab + MTX: Participants received rituximab 1000 mg IV and methylprednisolone 100 mg IV on Days 1 and 15. Participants should have been receiving a stable dose (for at least 12 weeks prior to Screening) of MTX 10-25 mg/week and a stable dose of folate (≥5 mg/week) given as either a single weekly dose or as divided daily doses (per investigator discretion). Participants who, in the opinion of the investigator, achieved a clinically relevant response (DAS28 score of ≥2.6) to the first course of treatment received one additional course of re-treatment with rituximab (2 IV infusions of rituximab 1000 mg [and methylprednisolone 100 mg] given 14 days apart), at any time between Week 24 and 48.
Arm/Group | Re-Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 77
percentage of participants
  With an AE | 68.8
  With a drug-related AE | 27.3
  With an acute infusion reaction | 13.0
  With AE leading to study drug discontinuation | 1.3
  With an SAE | 9.1
  With infections | 27.3
  With a serious infections | 2.6
  Who died | 0

3. Secondary Outcome: Percentage of Participants Meeting American College of Rheumatology (ACR) Response Criteria During the Initial Treatment Period
Description: ACR20/50/70, defined as ≥20 percent (%), 50%, or 70% improvement, respectively, compared to baseline in tender joint count (TJC) and swollen joint count (SJC), and 20%/50%/70% improvement in at least 3 of 5 additional ACR core set variables: Patient Assessment of Pain; Patient's Global Assessment of Disease Activity; Physician's Global Assessment of Disease Activity; Health Assessment Questionnaire - Disability Index (HAQ-DI); and an acute phase reactant (erythrocyte sedimentation rate [ESR] or C-Reactive Protein [CRP]). If CRP was missing or not done, then ESR was used.
Time Frame: Weeks 4, 12, 24, 36, and 48 of Initial treatment period
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
percentage of participants
  ACR20, Week 4 | 31.7
  ACR20, Week 12 | 50.0
  ACR20, Week 24 | 54.2
  ACR20, Week 36 | 25.0
  ACR20, Week 48 | 15.8
  ACR50, Week 4 | 5.8
  ACR50, Week 12 | 22.5
  ACR50, Week 24 | 25.0
  ACR50, Week 36 | 11.7
  ACR50, Week 48 | 9.2
  ACR70, Week 4 | 0
  ACR70, Week 12 | 4.2
  ACR70, Week 24 | 5.8
  ACR70, Week 36 | 5.8
  ACR70, Week 48 | 4.2
Statistical Analysis 1: Comparison: Initial Treatment Period: Rituximab + MTX; ACR20: Week 12 versus (vs) Week 4; Test type: Superiority or Other; p = 0.253, Regression, Logistic; Odds Ratio (OR) = 2.293
Statistical Analysis 2: Comparison: Initial Treatment Period: Rituximab + MTX; ACR20: Week 24 vs Week 4; Test type: Superiority or Other; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 3.019
Statistical Analysis 3: Comparison: Initial Treatment Period: Rituximab + MTX; ACR50: Week 12 vs Week 4; Test type: Superiority or Other; p = 0.023, Regression, Logistic; Odds Ratio (OR) = 5.552
Statistical Analysis 4: Comparison: Initial Treatment Period: Rituximab + MTX; ACR50: Week 24 vs. Week 4; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 6.861

4. Secondary Outcome: Percentage of Participants With Complete Clinical Response Per ACR Criteria During the Initial Treatment Period
Description: Complete clinical response was defined as having an ACR70 for at least 13 weeks.
Time Frame: Weeks 4, 12, 24, 36, and 48 of Initial treatment period
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
percentage of participants | 4.2

5. Secondary Outcome: Percentage of Participants Meeting ACR Response Criteria During the Re-treatment Period
Description: ACR20/50/70, defined as ≥20%, 50%, or 70% improvement, respectively, compared to baseline in TJC and SJC, and 20%/50%/70% improvement in at least 3 of 5 additional ACR core set variables: Patient Assessment of Pain; Patient's Global Assessment of Disease Activity; Physician's Global Assessment of Disease Activity; HAQ-DI; and an acute phase reactant (ESR or CRP). If CRP was missing or not done, then ESR was used.
Time Frame: Weeks 12 and 24 of Re-treatment period
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Re-Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 77
percentage of participants
  ACR20, Week 12 | 54.5
  ACR20, Week 24 | 58.4
  ACR50, Week 12 | 26.0
  ACR50, Week 24 | 28.6
  ACR70, Week 12 | 6.5
  ACR70, Week 24 | 9.1

6. Secondary Outcome: Percentage of Participants With Complete Clinical Response Per ACR Criteria During the Re-Treatment Period
Description: Complete clinical response was defined as having an ACR70 for at least 13 weeks.
Time Frame: Weeks 12 and 24 of Re-treatment period
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Re-Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 77
percentage of participants | 1.3

7. Secondary Outcome: Percentage of Participants Meeting European League Against Rheumatism (EULAR) Response Criteria During the Initial Treatment Period
Description: The EULAR response criteria were based on the assessment of disease activity using the DAS28. The EULAR response criteria included not only change in disease activity but current disease activity. To be classified as responders, participants had to have a significant change in DAS28 and a low current disease activity. There were 4 categories of EULAR response rates: good, moderate, good/moderate, and none. The DAS28 scoring used 4 core components: SJC, TJC, Patient's Global Assessment of Disease Activity, and ESR. The DAS28 has a continuous scale ranging from 0 to 9.4. The level of disease activity was interpreted as low (DAS28 score less than or equal to [≤]3.2), moderate (DAS28 score greater than [>]3.2 but ≤5.1), or high (DAS28 score >5.1). A DAS28 score <2.6 corresponded to a state of remission according to American Rheumatism Association criteria.
Time Frame: Weeks 4, 12, 24, 36, and 48 of Initial treatment period
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
percentage of participants
  Week 4: Good | 4.2
  Week 4: Moderate | 47.5
  Week 4: Good/Moderate | 51.7
  Week 4: None | 46.7
  Week 12: Good | 9.2
  Week 12: Moderate | 55.0
  Week 12: Good/Moderate | 64.2
  Week 12: None | 33.3
  Week 24: Good | 17.5
  Week 24: Moderate | 50.0
  Week 24: Good/Moderate | 67.5
  Week 24: None | 26.7
  Week 36: Good | 10.8
  Week 36: Moderate | 24.2
  Week 36: Good/Moderate | 35.0
  Week 36: None | 23.3
  Week 48: Good | 8.3
  Week 48: Moderate | 10.8
  Week 48: Good/Moderate | 19.2
  Week 48: None | 10.0
Statistical Analysis 1: Comparison: Initial Treatment Period: Rituximab + MTX; Good vs Moderate vs None: Week 12 vs Week 4; Test type: Superiority or Other; p = 0.667, Regression, Logistic; Odds Ratio (OR) = 2.099
Statistical Analysis 2: Comparison: Initial Treatment Period: Rituximab + MTX; Good vs Moderate vs None: Week 24 vs Week 4; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.589
Statistical Analysis 3: Comparison: Initial Treatment Period: Rituximab + MTX; Good/Moderate vs None: Week 12 vs Week 4; Test type: Superiority or Other; p = 0.440, Regression, Logistic; Odds Ratio (OR) = 2.138
Statistical Analysis 4: Comparison: Initial Treatment Period: Rituximab + MTX; Good/Moderate vs None: Week 24 vs Week 4; Test type: Superiority or Other; p = 0.012, Regression, Logistic; Odds Ratio (OR) = 3.009

8. Secondary Outcome: Percentage of Participants Meeting EULAR Response Criteria During the Re-Treatment Period
Description: The EULAR response criteria were based on the assessment of disease activity using the DAS28. The EULAR response criteria included not only change in disease activity but current disease activity. To be classified as responders, participants had to have a significant change in DAS28 and a low current disease activity. There were 4 categories of EULAR response rates: good, moderate, good/moderate, and none. The DAS28 scoring used 4 core components: SJC, TJC, Patient's Global Assessment of Disease Activity, and ESR. The DAS28 has a continuous scale ranging from 0 to 9.4. The level of disease activity was interpreted as low (DAS28 score ≤3.2), moderate (DAS28 score >3.2 but ≤5.1), or high (DAS28 score >5.1). A DAS28 score <2.6 corresponded to a state of remission according to American Rheumatism Association criteria.
Time Frame: Weeks 12 and 24 of Re-treatment period
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Re-Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 77
percentage of participants
  Week 12: Good | 20.8
  Week 12: Moderate | 53.2
  Week 12: Good/Moderate | 74.0
  Week 12: None | 22.1
  Week 24: Good | 19.5
  Week 24: Moderate | 48.1
  Week 24: Good/Moderate | 67.5
  Week 24: None | 26.0

9. Secondary Outcome: Change From Baseline in DAS28 During the Initial Treatment Period
Description: The DAS28 scoring used 4 core components: SJC, TJC, Patient's Global Assessment of Disease Activity, and ESR. The DAS28 has a continuous scale ranging from 0 to 9.4. The level of disease activity was interpreted as low (DAS28 score ≤3.2), moderate (DAS28 score >3.2 but ≤5.1), or high (DAS28 score >5.1). A DAS28 score <2.6 corresponded to a state of remission according to American Rheumatism Association criteria. A change of 1.2 units in DAS28 in an individual participant was considered a significant change.
Time Frame: Weeks 4, 12, 24, 36, and 48 of Initial treatment period
Population: ITT Population; n (number) = number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 117
scores on a scale
  Baseline (n=117) | 6.4 (1.1)
  Change at Week 4 (n=112) | -1.1 (0.8)
  Change at Week 12 (n=108) | -1.7 (1.2)
  Change at Week 24 (n=105) | -2.0 (1.2)
  Change at Week 36 (n=66) | -1.7 (1.7)
  Change at Week 48 (n=33) | -2.1 (1.6)
Statistical Analysis 1: Comparison: Initial Treatment Period: Rituximab + MTX; Week 4; Test type: Superiority or Other; p < 0.001, t-test, 1 sided
Statistical Analysis 2: Comparison: Initial Treatment Period: Rituximab + MTX; Week 12; Test type: Superiority or Other; p < 0.001, t-test, 1 sided
Statistical Analysis 3: Comparison: Initial Treatment Period: Rituximab + MTX; Week 24; Test type: Superiority or Other; p < 0.001, t-test, 1 sided
Statistical Analysis 4: Comparison: Initial Treatment Period: Rituximab + MTX; Week 36; Test type: Superiority or Other; p < 0.001, t-test, 1 sided
Statistical Analysis 5: Comparison: Initial Treatment Period: Rituximab + MTX; Week 48; Test type: Superiority or Other; p < 0.001, t-test, 1 sided

10. Secondary Outcome: Change From Baseline in DAS28 During the Re-Treatment Period
Description: The DAS28 scoring used 4 core components: SJC, TJC, Patient Global Assessment of Disease Activity, and ESR. The DAS28 has a continuous scale ranging from 0 to 9.4. The level of disease activity was interpreted as low (DAS28 score ≤3.2), moderate (DAS28 score >3.2 but ≤5.1), or high (DAS28 score >5.1). A DAS28 score <2.6 corresponded to a state of remission according to American Rheumatism Association criteria. A change of 1.2 units in DAS28 in an individual participant was considered a significant change.
Time Frame: Weeks 12 and 24 of Re-treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Re-Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 117
scores on a scale
  Baseline (n=117) | 6.4 (1.1)
  Change at Week 12 (n=70) | -2.3 (1.3)
  Change at Week 24 (n=65) | -2.2 (1.4)

11. Secondary Outcome: Change From Baseline in SJC During the Initial Treatment Period
Description: Joints assessed for swelling consisted of shoulders, elbows, wrists, interphalangeal (digit 1), distal interphalangeal joints (digits 2-5), proximal interphalangeal joints (digits 2-5), metacarpophalangeal joints (digits 1-5), and knees.
Time Frame: Weeks 4, 12, 24, 36, and 48 of Initial treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 117
swollen joints
  Baseline (n=117) | 13.7 (5.33)
  Change at Week 4 (n=115) | -3.6 (4.45)
  Change at Week 12 (n=113) | -5.7 (4.97)
  Change at Week 24 (n=106) | -7.1 (5.66)
  Change at Week 36 (n=67) | -5.6 (6.50)
  Change at Week 48 (n=33) | -7.7 (5.56)
Statistical Analysis 1: Comparison: Initial Treatment Period: Rituximab + MTX; Baseline vs Week 24; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed-Rank test

12. Secondary Outcome: Change From Baseline in SJC During the Re-Treatment Period
Description: as for outcome 11
Time Frame: Weeks 12 and 24 of Re-treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given vist.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 117
swollen joints
  Baseline (n=117) | 13.7 (5.33)
  Change at Week 12 (n=71) | -7.6 (6.07)
  Change at Week 24 (n=69) | -7.7 (5.43)

13. Secondary Outcome: Change From Baseline in TJC During the Initial Treatment Period
Description: as for outcome 11
Time Frame: Weeks 4, 12, 24, 36, and 48 of Initial treatment period
Population: ITT Population; n=number of participants assessed for the specific parameter at a given visit.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 117
tender joints
  Baseline (n=117) | 16.1 (6.62)
  Change at Week 4 (n=115) | -6.3 (5.95)
  Change at Week 12 (n=113) | -7.8 (6.68)
  Change at Week 24 (n=106) | -9.0 (6.42)
  Change at Week 36 (n=67) | -7.4 (8.35)
  Change at Week 48 (n=33) | -7.8 (8.31)
Statistical Analysis 1: Comparison: Initial Treatment Period: Rituximab + MTX; Baseline vs Week 24; Test type: Superiority or Other; p < 0.001, t-test, 1 sided

14. Secondary Outcome: Change From Baseline in TJC During the Re-Treatment Period
Description: as for outcome 11
Time Frame: Weeks 12 and 24 of Re-treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Re-Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 117
tender joints
  Baseline (n=117) | 16.1 (6.62)
  Change at Week 12 (n=71) | -9.4 (7.54)
  Change at Week 24 (n=69) | -9.7 (6.92)

15. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity During the Initial Treatment Period
Description: Physician Global Assessment of Disease Activity was measured using a 100-mm visual analog scale (VAS) where the extreme left end of the line was 0 = no disease activity and the extreme right end of the line was 100 = maximum disease activity. The physician marked the line and the distance from the left edge was measured in mm.
Time Frame: Weeks 4, 12, 24, 36, and 48 of Initial treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
mm
  Baseline (n=120) | 68.6 (17.34)
  Change at Week 4 (n=117) | -22.0 (21.67)
  Change at Week 12 (n=116) | -31.4 (24.28)
  Change at Week 24 (n=109) | -35.1 (24.45)
  Change at Week 36 (n=68) | -28.6 (28.68)
  Change at Week 48 (n=34) | -35.9 (25.18)
Statistical Analysis 1: Comparison: Initial Treatment Period: Rituximab + MTX; Baseline vs Week 24; Test type: Superiority or Other; p < 0.001, t-test, 1 sided

16. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity During the Re-Treatment Period
Description: Physician Global Assessment of Disease Activity was measured using a 100-mm VAS where the extreme left end of the line was 0 = no disease activity and the extreme right end of the line was 100 = maximum disease activity. The physician marked the line and the distance from the left edge was measured in mm.
Time Frame: Weeks 12 and 24 of Re-treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Re-Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
mm
  Baseline (n=120) | 68.6 (17.34)
  Change at Week 12 (n=73) | -35.5 (25.95)
  Change at Week 24 (n=69) | -41.5 (24.43)

17. Secondary Outcome: Change From Baseline in Patient Global Assessment of Disease Activity Score During the Initial Treatment Period
Description: Patient Global Assessment of Disease Activity was measured using a 100-mm VAS where the extreme left end of the line was 0 = no disease activity and the extreme right end of the line was 100 = maximum disease activity. The participant was asked to marked the line and the distance from the left edge was measured in mm.
Time Frame: Weeks 4, 12, 24, 36, and 48 of Initial treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
mm
  Baseline (n=120) | 67.5 (22.73)
  Change at Week 4 (n=117) | -19.7 (21.50)
  Change at Week 12 (n=116) | -26.3 (26.84)
  Change at Week 24 (n=109) | -29.2 (25.72)
  Change at Week 36 (n=68) | -23.8 (30.42)
  Change at Week 48 (n=34) | -28.5 (22.92)
Statistical Analysis 1: Comparison: Initial Treatment Period: Rituximab + MTX; Baseline vs Week 24; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test

18. Secondary Outcome: Change From Baseline in Patient Global Assessment of Disease Activity During the Re-Treatment Period
Description: as for outcome 17
Time Frame: Weeks 12 and 24 of Re-treatment period and Week 4 after last maintenance
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Re-Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
mm
  Baseline (n=120) | 67.5 (22.73)
  Change at Week 12 (n=72) | -32.6 (29.20)
  Change at Week 24 (n=72) | -30.7 (28.70)

19. Secondary Outcome: Change From Baseline in Patient Global Assessment of Pain During the Initial Treatment Period
Description: Patient Global Assessment of Pain was measured using a 100-mm VAS where the extreme left end of the line was 0 = no pain and the extreme right end of the line was 100 = unbearable pain. The participant was asked to mark the line and the distance from the left edge was measured in mm.
Time Frame: Weeks 4, 12, 24, 36, and 48 of Initial treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
mm
  Baseline (n=120) | 60.2 (22.85)
  Change at Week 4 (n=117) | -17.5 (21.80)
  Change at Week 12 (n=113) | -24.0 (25.31)
  Change at Week 24 (n=108) | -25.7 (25.40)
  Change at Week 36 (n=68) | -18.0 (29.18)
  Change at Week 48 (n=33) | -22.6 (20.07)
Statistical Analysis 1: Comparison: Initial Treatment Period: Rituximab + MTX; Baseline vs Week 24; Test type: Superiority or Other; p < 0.001, t-test, 1 sided

20. Secondary Outcome: Change From Baseline in Patient Global Assessment of Pain During the Re-Treatment Period
Description: as for outcome 19
Time Frame: Weeks 12 and 24 of Re-treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Re-Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
mm
  Baseline (n=120) | 60.2 (22.85)
  Change at Week 12 (n=72) | -28.3 (28.02)
  Change at Week 24 (n=72) | -26.6 (27.61)

21. Secondary Outcome: Change From Baseline HAQ-DI Score During the Initial Treatment Period
Description: HAQ-DI: 20 questions, 8 categories of functioning: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common usual activities. Participants report amount of difficulty in performing 2-3 specific subcategory items. Difficulty score is from 0 to 3 (0 = without any difficulty; 1 = with some difficulty; 2 = with much difficulty; and 3 = unable to do). The highest component score in each of the 8 categories determined the score for that category, unless aids, devices, and/or help from another person were required which = a score of 2 (unless already 2 or 3). The 8 category scores were averaged into overall HAQ-DI score ranging from 0 to 3 (0 to 1 = mild to moderate difficulty; 1 to 2 = moderate to severe disability; and 2 to 3 = severe to very severe disability). HAQ-DI not computed if > 2 categories were missing.
Time Frame: Weeks 4, 12, 24, 36, and 48 of Initial treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
scores on a scale
  Baseline (n=120) | 1.7 (0.57)
  Change at Week 4 (n=117) | -0.2 (0.36)
  Change at Week 12 (n=116) | -0.3 (0.46)
  Change at Week 24 (n=108) | -0.4 (0.48)
  Change at Week 36 (n=68) | -0.3 (0.53)
  Change at Week 48 (n=34) | -0.4 (0.56)
Statistical Analysis 1: Comparison: Initial Treatment Period: Rituximab + MTX; Baseline vs Week 24; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test

22. Secondary Outcome: Change From Baseline HAQ-DI Score During the Re-Treatment Period
Description: HAQ-DI: 20 questions, 8 categories of functioning: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common usual activities. Participants report amount of difficulty in performing 2-3 specific subcategory items. Difficulty score is from 0 to 3 (0 = without any difficulty; 1 = with some difficulty; 2 = with much difficulty; and 3 = unable to do). The highest component score in each of the 8 categories determines the score for that category, unless aids, devices, and/or help from another person were required which = a score of 2 (unless already 2 or 3). The 8 category scores were averaged into overall HAQ-DI score ranging from 0 to 3 (0 to 1 = mild to moderate difficulty; 1 to 2 = moderate to severe disability; and 2 to 3 = severe to very severe disability). HAQ-DI not computed if >2 categories were missing.
Time Frame: Weeks 12 and 24 of Re-treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Re-Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
scores on a scale
  Baseline (n=120) | 1.7 (0.57)
  Change at Week 12 (n=73) | -0.5 (0.60)
  Change at Week 24 (n=72) | -0.5 (0.62)

23. Secondary Outcome: Change From Baseline in ESR During the Initial Treatment Period
Description: ESR was measured in mm/hour and was used to determine the acute phase response. Lower ESR values indicate reduction in disease activity; normal reference range: 0-20 mm/hr.
Time Frame: Weeks 4, 12, 24, 36, and 48 of Initial treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
mm/hr
  Baseline (n=120) | 37.0 (27.84)
  Change at Week 4 (n=112) | -4.5 (13.57)
  Change at Week 12 (n=112) | -11.3 (20.60)
  Change at Week 24 (n=107) | -16.0 (20.36)
  Change at Week 36 (n=68) | -9.2 (22.29)
  Change at Week 48 (n=34) | -12.0 (17.93)
Statistical Analysis 1: Comparison: Initial Treatment Period: Rituximab + MTX; Baseline vs Week 24; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test

24. Secondary Outcome: Change From Baseline in ESR During the Re-Treatment Period
Description: as for outcome 23
Time Frame: Weeks 12 and 24 of Re-treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Re-Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
mm/hr
  Baseline (n=120) | 37.0 (27.84)
  Change at Week 12 (n=73) | -17.9 (22.07)
  Change at Week 24 (n=67) | -18.7 (23.05)

25. Secondary Outcome: Change From Baseline in CRP During the Initial Treatment Period
Description: CRP levels were measured in milligrams/liter (mg/L) and were used to determine the acute phase response. A reduction in CRP levels is considered an improvement; normal reference range ≤10 mg/L.
Time Frame: Weeks 4, 12, 24, 36, and 48 of Initial treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 119
mg/L
  Baseline (n=119) | 25.6 (28.87)
  Change at Week 4 (n=110) | -7.9 (17.44)
  Change at Week 12 (n=113) | -11.9 (31.97)
  Change at Week 24 (n=108) | -16.1 (24.82)
  Change at Week 36 (n=67) | -9.1 (25.74)
  Change at Week 48 (n=34) | -7.6 (27.06)
Statistical Analysis 1: Comparison: Initial Treatment Period: Rituximab + MTX; Baseline vs Week 24; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test

26. Secondary Outcome: Change From Baseline CRP During the Re-Treatment Period
Description: CRP levels were measured in mg/L and were used to determine the acute phase response. A reduction in CRP levels is considered an improvement; normal reference range ≤10 mg/L.
Time Frame: Weeks 12 and 24 of Re-treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Re-Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 119
mg/L
  Baseline (n=119) | 25.6 (28.87)
  Change at Week 12 (n=70) | -16.9 (27.15)
  Change at Week 24 (n=67) | -15.3 (26.62)

27. Secondary Outcome: Percentage of Participants With Disease Remission According to DAS28 in the Initial Treatment Period
Description: The DAS28 scoring used 4 core components: SJC, TJC, Patient's Global Assessment of Disease Activity, and ESR. The DAS28 has a continuous scale ranging from 0 to 9.4. The level of disease activity was interpreted as low (DAS28 score ≤3.2), moderate (DAS28 score >3.2 but ≤5.1), or high (DAS28 score >5.1). A DAS28 score ≤2.6 corresponded to a state of remission according to American Rheumatism Association criteria.
Time Frame: Weeks 4, 12, 24, 36, and 48 of Initial treatment period
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
percentage of participants
  Week 4 | 0.8
  Week 12 | 5.0
  Week 24 | 5.8
  Week 36 | 5.8
  Week 48 | 5.8

28. Secondary Outcome: Percentage of Participants With Disease Remission According to DAS28 in the Re-Treatment Period
Description: as for outcome 27
Time Frame: Weeks 12 and 24 of Re-treatment period
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Re-Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 77
percentage of participants
  Week 12 | 5.0
  Week 24 | 4.2

29. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Total Score During the Initial Treatment Period
Description: Participant fatigue was evaluated using the FACIT-F scale, a 13-item questionnaire in which the participants were requested to score each item on a 5-point scale. The FACIT-F scores ranged from 0 to 52, with higher scores representing less fatigue. Score changes of 4 points or more were considered clinically meaningful. The total score was a summation of all 13 items, where 2 of the positive items (I have energy; I am able to do my usual activities) were reversed for scoring.
Time Frame: Weeks 4, 12, 24, 36, and 48 of Initial treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Initial Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
scores on a scale
  Baseline (n=120) | 28.9 (10.22)
  Change at Week 4 (n=116) | -5.4 (8.19)
  Change at Week 12 (n=116) | -7.3 (10.38)
  Change at Week 24 (n=108) | -9.1 (9.90)
  Change at Week 36 (n=68) | -8.6 (11.71)
  Change at Week 48 (n=34) | -10.9 (10.68)
Statistical Analysis 1: Comparison: Initial Treatment Period: Rituximab + MTX; Baseline vs Week 12; Test type: Superiority or Other; p < 0.001, t-test, 1 sided
Statistical Analysis 2: Comparison: Initial Treatment Period: Rituximab + MTX; Baseline vs Week 24; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank test

30. Secondary Outcome: Change From Baseline in FACIT-F Total Score During the Re-Treatment Period
Description: as for outcome 29
Time Frame: Weeks 12 and 24 of Re-treatment period
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Re-Treatment Period: Rituximab + MTX
Number analyzed (Participants) | 120
scores on a scale
  Baseline (n=120) | 28.9 (10.22)
  Change at Week 12 (n=73) | -8.3 (12.64)
  Change at Week 24 (n=72) | -8.9 (11.72)

ADVERSE EVENTS:
Time Frame: Reporting period began after written informed consent was obtained and ended 48 weeks after therapy was initiated or 24 weeks after re-treatment had occurred.
Description: Participants removed from therapy and entered into the Safety Follow-up period were followed for AEs for an additional 24 weeks after the cessation of therapy, whether considered treatment-related or not. Nonserious adverse events presented in this record include all adverse events reported during the study, not just nonserious events.
Groups:
- Initial Treatment: Rituximab + MTX: Participants received rituximab 1000 mg IV and methylprednisolone 100 mg IV on Days 1 and 15. Participants should have been receiving a stable dose (for at least 12 weeks prior to Screening) of MTX 10-25 mg/week and a stable dose of folate (≥5 mg/week) given as either a single weekly dose or as divided daily doses (per investigator discretion).
- Re-treatment: Rituximab + MTX: Participants received rituximab 1000 mg IV and methylprednisolone 100 mg IV on Days 1 and 15. Participants should have been receiving a stable dose (for at least 12 weeks prior to Screening) of MTX 10-25 mg/week and a stable dose of folate (≥5 mg/week) given as either a single weekly dose or as divided daily doses (per investigator discretion). Participants who, in the opinion of the investigator, achieved a clinically relevant response (DAS28 score of ≥2.6) to the first course of treatment received one additional course of re-treatment with rituximab (2 IV infusions of rituximab 1000 mg [and methylprednisolone 100 mg] given 14 days apart), at any time between Week 24 and 48.
Arm/Group | Initial Treatment: Rituximab + MTX | Re-treatment: Rituximab + MTX
Serious Adverse Events (participants affected / at risk) | 12/120 | 7/77
Other Adverse Events (participants affected / at risk) | 102/120 | 53/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Treatment: Rituximab + MTX (N=120) | Re-treatment: Rituximab + MTX (N=77)
Labyrinthitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Breast cellulitis (Infections and infestations) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Treatment: Rituximab + MTX (N=120) | Re-treatment: Rituximab + MTX (N=77)
Nasopharyngitis (Infections and infestations) | 13 | 8
Upper respiratory tract infection (Infections and infestations) | 7 | 3
Urinary tract infection (Infections and infestations) | 9 | 3
Sinusitis (Infections and infestations) | 6 | 1
Bronchitis (Infections and infestations) | 6 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 20 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 3
Nausea (Gastrointestinal disorders) | 17 | 9
Diarrhoea (Gastrointestinal disorders) | 7 | 4
Vomiting (Gastrointestinal disorders) | 7 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 4
Headache (Nervous system disorders) | 14 | 6
Dizziness (Nervous system disorders) | 9 | 3
Fatigue (General disorders) | 10 | 1
Oedema peripheral (General disorders) | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 2
Flushing (Vascular disorders) | 7 | 0

LIMITATIONS AND CAVEATS:
Nonserious adverse events presented in this record include all adverse events reported during the study, not just nonserious events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.